CLINICAL TRIAL: NCT01094262
Title: A Randomized, Double-Blind, Placebo- and Active-Controlled Study to Evaluate the Efficacy, Safety and Tolerability of JNJ-42160443 as Monotherapy in Subjects With Moderate to Severe, Chronic Knee Pain From Osteoarthritis
Brief Title: A Safety and Tolerability Study of JNJ-42160443 in Patients With Moderate to Severe, Chronic Knee Pain From Osteoarthritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Logistic reasons associated with the FDA-imposed clinical hold.
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR017092; 42160443-PAI2006 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.); 2009-016831-36 (EudraCT Number)
Record Dates: First submitted 2010-03-25; First posted 2010-03-26 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Osteoarthritis; Osteoarthritis, Knee; Pain; Arthralgia; Joint Pain
Keywords: Osteoarthritis pain of the knee; Osteoarthritis; Osteoarthritis, Knee; Pain; Arthralgia; Joint Pain; JNJ-42160443
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee; Pain; Arthralgia | interventions — fulranumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (4):
- JNJ-42160443 (lower dose) (Experimental)
  Interventions: Drug: JNJ-42160443
- JNJ-42160443 (higher dose) (Experimental)
  Interventions: Drug: JNJ-42160443
- Oxycodone CR (standard pain medication) (Active Comparator)
  Interventions: Drug: Oxycodone CR (standard pain medication)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxycodone CR (standard pain medication) — Oxycodone CR: Type=exact number, unit=mg, number= 10-50, form=capsule, route=oral use and Placebo: Form=solution for injection, route=Subcutaneous use. Oxycodone CR capsule twice a day for 16 weeks and one placebo injection every 4 weeks for 16 weeks.
  Arms: Oxycodone CR (standard pain medication)
Drug: JNJ-42160443 — JNJ-42160443: Type=exact number, unit=mg, number= 3, form=solution for injection, route=Subcutaneous use and Placebo: Form=capsule, route=Oral use. One injection of JNJ-42160443 every 4 weeks and a placebo capsule twice a day for 16 weeks.
  Arms: JNJ-42160443 (lower dose)
Drug: JNJ-42160443 — JNJ-42160443: Type=exact number, unit=mg, number= 9, form=solution for injection, route=Subcutaneous use and Placebo: Form=capsule, route=Oral use. One injection of JNJ-42160443 every 4 weeks and a placebo capsule twice a day for 16 weeks.
  Arms: JNJ-42160443 (higher dose)
Drug: Placebo — Form=solution for injection, route=Subcutaneous use and Form=capsule, route=Oral use. One placebo injection every 4 weeks and a placebo capsule twice a day for 16 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate pain relief, safety, and tolerability of a new treatment (JNJ-42160443) for moderate to severe pain of osteoarthritis of the knee in comparison to a standard pain treatment and placebo.

DETAILED DESCRIPTION:
This is a double-blind (neither the physician nor the patient knows the name of the assigned drug) study evaluating pain relief, safety, and tolerability of a new treatment (JNJ-42160443) for moderate to severe pain of osteoarthritis of the knee in comparison to a standard pain treatment and placebo. The study will last for about 42 weeks. Patients will receive treatment for 16 weeks. Patients who qualify for the study based on their level of pain as well as other factors will receive one of the 4 possible treatments as determined by chance. Before entering the study, patients must stop using their present pain medication. During the study, patients will answer questions about their pain, side effects, and have tests performed to monitor their physical condition. The main purpose of the study is to compare pain relief with JNJ-42160443 to that of a standard pain treatment or placebo. After the treatment period, patients can return to taking the pain medication that they used before the start of the study, and their physical condition will continue to be monitored. JNJ 42160443 10 mg/mL will be provided for use in the study. Patients will receive 1 of 4 treatments for 16 weeks (wks): lower dosage of JNJ 42160443 by subcutaneous (under the skin) (SC) injection once every 4 wks + Placebo (P) capsule orally (by mouth) (PO) 2x/day, higher dosage of JNJ 42160443 by SC injection once every 4 wks + P capsule PO 2x/day, standard pain medication capsule PO 2x/day + P by SC injection once every 4 wks, or P capsule PO 2x/day + P by SC injection once every 4 wks.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of osteoarthritis of the knee
* Have moderate to severe pain based on a trial questionnaire
* Must be on a stable dose of pain medication for 4 weeks before entering the trial
* Medically stable condition

Exclusion Criteria:

* History of joint replacement surgery in the affected joint or planned surgery involving the affected joint during the trial
* Diabetes mellitus
* Uncontrolled cardiovascular disease or hypertension
* Previous treatment with another investigational NGF inhibitor therapy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2010-04-20 (Actual); Primary Completion 2011-07-01 (Actual); Study Completion 2011-07-01 (Actual)

PRIMARY OUTCOMES:
Change in the average daily pain intensity | From Baseline to Week 13 (ie, after 12 weeks of treatment)

SECONDARY OUTCOMES:
Western Ontario and McMaster Osteoarthritis Index (WOMAC 3.1) subscales scores | 12 weeks
  The WOMAC 3.1 is a multi-dimensional, osteoarthritis specific questionnaire designed to assess clinically important symptoms of the hip and/or knee.
Patient Global Assessment (PGA) scale score | 12 weeks
  The PGA is a single item that the patient completes to indicate their perception of their osteoarthritis status, on an 11-point numerical rating scale from 0 (Very Good) to 10 (Very Bad).

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (44):
- United States (36):
  - Tucson, Arizona
  - Carmichael, California
  - Pismo Beach, California
  - Clearwater, Florida
  - Hallandale, Florida
  - Oldsmar, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Marietta, Georgia
  - Perry, Georgia
  - Woodstock, Georgia
  - Boise, Idaho
  - Eagle, Idaho
  - Avon, Indiana
  - Evansville, Indiana
  - Baton Rouge, Louisiana
  - Mandeville, Louisiana
  - Metairie, Louisiana
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Watertown, Massachusetts
  - St Louis, Missouri
  - Omaha, Nebraska
  - Mamaroneck, New York
  - Williamsville, New York
  - Greenville, North Carolina
  - Raleigh, North Carolina
  - Kettering, Ohio
  - Oklahoma City, Oklahoma
  - Collegeville, Pennsylvania
  - Duncansville, Pennsylvania
  - Grapevine, Texas
  - Lubbock, Texas
  - Odessa, Texas
  - Richardson, Texas
  - San Antonio, Texas
- Canada (8):
  - Corunna, Ontario
  - Greater Sudbury, Ontario
  - London, Ontario
  - Newmarket, Ontario
  - Sarnia, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec

REFERENCES:
- [Derived] Mayorga AJ, Wang S, Kelly KM, Thipphawong J. Efficacy and safety of fulranumab as monotherapy in patients with moderate to severe, chronic knee pain of primary osteoarthritis: a randomised, placebo- and active-controlled trial. Int J Clin Pract. 2016 Jun;70(6):493-505. doi: 10.1111/ijcp.12807. PMID 27238963